CLINICAL TRIAL: NCT05689892
Title: Impact of a Shared Decision Making Intervention in Paediatric Inflammatory Bowel Disease Therapeutic Decision-making
Brief Title: Shared Decision Making in Paediatric Inflammatory Bowel Disease
Acronym: SDM-IBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Eileen Crowley, Physician, Assistant Professor, London Health Sciences Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12069
Record Dates: First submitted 2022-12-13; First posted 2023-01-19 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; IBD
Keywords: decisional conflict; shared decision making; SDM; decisional regret; biologics; biologic therapy; pediatric IBD; pIBD
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants who have been diagnosed with IBD and are recommended a new biologic therapy will be recruited to this arm. Participants and their families will be referred to a decision coach (DC), who will provide support in gaining knowledge of treatment and care options. They will also be given decision aids (DA) as outlined in the study description.
  Interventions: Other: Decision Coach Sessions
- Comparator group (No Intervention): Participants who have been recommended a new biologic therapy within the last 12 months and have commenced treatment will be recruited to this arm.

INTERVENTIONS:
Other: Decision Coach Sessions — Participants in the intervention group and their families will be referred to the DC to meet independently and discuss recommended treatment pathways.
  Multiple sessions may be necessary until a final decision is reached. All SDM consults will be done virtually using a secure videoconferencing platform. The Ottawa Family Decision Guide will be used to facilitate the discussion. A DA will be provided to the study participants in the form of information cards containing information about different treatment options in pediatric IBD. This includes administration schedule, side effects, risk of cancer, among others. The DA has been developed and provided by the Cincinnati Children's Hospital Medical Center and adapted to the Canadian setting with electronic version by this research group with approval from the authors.
  Other Names: DC sessions
  Arms: Intervention group

SUMMARY:
The goal of this mixed-methods prospective cohort study is to assess the impact of shared decision-making (SDM) on newly diagnosed pediatric inflammatory bowel disease (IBD) patients and their families. Patient and familial decisional conflict regarding the choice and course of treatment is shown to be high, especially for the newer class of IBD treatments called biologic agents. SDM intervention comprises of coaching with a decision coach (DC) on all aspects of treatment and care, along with educational decision aids (DA) provided and adapted from Cincinnati Children's Hospital Medical Center.

The main aims of this study are:

1. to determine if SDM intervention has an impact on patient and parental decision making in pediatric IBD treatments, mainly by assessing decisional conflict and decision satisfaction/regret.
2. to adapt and assess the acceptability of DA in a Canadian academic center.

Participants who have been recommended a new biologic as part of their clinical care for IBD will be recruited to the SDM intervention group. The participants will have DC sessions until a final treatment decision is made, will be given DAs, and will be followed by baseline and post-intervention surveys to assess decisional conflict and satisfaction/regret.

The comparator group will include participants who have been recommended and have commenced a new biologic within the last 12 months.

Outcome metrics will evaluate the impact on parental and patient decisional conflict following SDM intervention, and decisional satisfaction/regret 6-12 months from therapy start.

DETAILED DESCRIPTION:
Rationale Patient and family-centered care has become prevalent in the last few decades, recognizing the pivotal role of patients and their families in the decision-making process. Partnering with the healthcare team improves decision making, reduces uncertainty and conflicts that often accompany complex decisions, potentially leading to better outcomes for the patient and family. This shared decision-making (SDM) employs decision aids (DA) and/or an impartial Decision Coach (DC) as a foundation to help patients be actively involved in their care and ensure the best outcomes.

A group of chronic diseases with complicated prognoses and poorly understood pathophysiology, Inflammatory Bowel Disease (IBD) has shown increasing incidence in children. Long-term therapy is required to maintain remission. About 60% of patients undergo biologic therapy, many needing a change of therapy or surgery due to failed initial induction. The availability of multiple biologic therapies for paediatric IBD (pIBD), each with risks, benefits and side effects, modes of administrations, dosing and insurance coverage issues, frequently overwhelms patients and parents when deciding on initial therapies. Delays in the decision process may also result in further complications and reduced steroid-free remission rates.

This project will investigate the impact of SDM on familial stress, decisional confidence and decisional regret of pIBD patients and their families. Expected outcomes are a change in decisional conflict and regret, leading to improved efficiency and quality of care supporting the need for this approach in all healthcare settings.

Aims and Hypothesis The aim of this pilot study is to evaluate whether an SDM intervention has an impact on patient and parental decision making in pIBD treatments, focusing on the constructs of decisional conflict and decision satisfaction/regret. The secondary aim is to adapt and assess the acceptability of the DA in a Canadian academic center.

The investigators hypothesize that: 1) Parents and adolescent patients will experience reduced conflict post-decision because of the SDM intervention. 2) The SDM intervention will reduce decisional regret 6 months after the treatment decision. 3) The DA will be accepted and have a positive effect on patient and parent preparation for decision making. 4) Patients and parents will be satisfied with the DC session.

Study design and methods This is a mixed methods prospective cohort and case-control pilot study. Recruitment: 75 parents of pIBD patients will be recruited in the intervention and comparator groups each over 2 years' time. New biologic therapy patients will be in the intervention group, those who have been on a biologic within the last 12 months in the comparator group. Patients referred to the SDM program at Children's Hospital, London Health Sciences Centre (LHSC) by the clinicians (Dr. Eileen Crowley, Dr. Dhandapani Ashok, and Dr. Kevin Bax) will be prospectively screened for enrollment and initially approached for the study by the clinicians. Interested patients will be provided letters of information and consent (assent if applicable - in the instance participants are unable to provide consent, since the population includes children and adolescents) by the clinicians or the research team prior to the session(s) with the DC. Participation in the study is voluntary and will not impact the clinical SDM process.

SDM Intervention: Intervention group families will be referred to the DC for independent virtual session(s) to discuss recommended treatment plans facilitated by the Ottawa Family Decision Guide. Multiple meetings may be necessary until a final decision is made. All SDM consults will be done virtually using a secure videoconferencing platform. The Ottawa Family Decision Guide will be used to facilitate the discussion. A DA will be provided to the study participants in the form of information cards containing information about different treatment options in pediatric IBD. This includes administration schedule, side effects, risk of cancer, among others. Sessions with the Decision Coach and the DAs provided will work in tandem to provide the best outcome for the patient and their family. The DA has been developed and provided by the Cincinnati Children's Hospital Medical Center and adapted to the Canadian setting with electronic version by this research group with approval from the authors.

Study procedures: Patient characteristics and clinical outcome data will be collected from medical charts. All information will be deidentified and anonymous, complying with the requirements for the protection of patient privacy and confidentiality. Intervention group participants will complete the baseline survey prior to any consultations. Validated SDM questionnaires will be applied during and post decision visit, as is part of the clinical program, with baseline questionnaires at first visit. Decisional regret will be assessed 6 months after therapy start. The validated questionnaires are:

1. SURE (Sure of myself; Understand information; Risk-benefit ratio; Encouragement) questionnaire and 16 item Decisional Conflict Scale pre/post SDM intervention,
2. Preparation for Decision Making Scale: acceptability and effect of DA following the intervention,
3. Decision Coach Questionnaire: acceptability of the DC session post intervention,
4. Decisional Regret Scale: distress or remorse after the treatment decision

Statistical analysis: Summary statistics will employ medians and interquartile ranges for continuous variables or means and standard deviations when appropriate. Frequencies with proportions will be used for categorical variables. A Wilcoxon signed-rank test will be used to measure change in decisional conflict pre- and post-intervention. Mann-Whitney U tests will be used to measure differences between intervention and comparator groups. SPSS v.27 (IBM Corp., Armonk, NY, USA) will be used for all analyses, and p-values <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking substitute decision makers and adolescent patients (age 13-17.99 years) with IBD that are recommended a new biologic therapy.
* English-speaking substitute decision makers and adolescent patients (age 13-17.99 years) with IBD that have started a new biologic therapy within the last 6 to 12 months, without SDM intervention.

Exclusion Criteria:

* patient over age 18
* non-English speakers
* acute medical instability or any known major mental illness in parent or adolescent patient

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on the16-item Decisional Conflict Scale (DCS) test to immediately after the Shared Decision Making intervention | baseline (before SDM intervention), immediately after the final SDM session
  The Decisional Conflict Scale is a 16-item measure that captures uncertainty in making choices related to health, the factors contributing to this uncertainty, and an individual's self-perceived satisfaction in the decision. The scale ranges from 0 (no decisional conflict) to 100 (extremely high decisional conflict).
  A Wilcoxon signed-rank test will be used to measure the change in test score. Mann-Whitney U tests will be used to measure differences between intervention and comparator groups. p-values < 0.05 will be considered statistically significant.
  Improvements in the test score by an effect size of 0.4 or more will determine the success of the study.
Change from baseline on the 4-item SURE (Sure of myself; Understand Information; Risk-benefit ratio; Encouragement) screening test to immediately after the Shared Decision Making intervention | baseline (before SDM intervention), immediately after the final SDM session
  The SURE Test is a screening test for the Decisional Conflict Scale (DCS) intended for use in everyday clinical practice. It can indicate the probability that a patient experiences clinically significant decisional conflict. Total scores range from 0 (extreme decisional conflict) to 4 (no decisional conflict).
  A Wilcoxon signed-rank test will be used to measure the change in test score. Mann-Whitney U tests will be used to measure differences between intervention and comparator groups. p-values < 0.05 will be considered statistically significant.
  An improvement of 4-point test score will determine the success of the study.
Change from baseline on the Decision Coach Questionnaire to immediately after the Shared Decision Making intervention | baseline (before SDM intervention), immediately after the final SDM session
  The Decision Coach Questionnaire is a validated SDM questionnaire to assess the acceptability and effect of decision coaching and decision aids.
  A Wilcoxon signed-rank test will be used to measure the change in test score. Mann-Whitney U tests will be used to measure differences between intervention and comparator groups. p-values < 0.05 will be considered statistically significant.
  An improvement of the mean Preparation for Decision Making score being above 3.8 (or 70) will determine the success of the study.

SECONDARY OUTCOMES:
Reduced decisional regret at 6-12 months after therapy start in the intervention group | baseline (before SDM intervention), 6-12 months after the final SDM session
  The DRS is a five-item, self-report scale to evaluate decisional regret. Items are scored on five-point Likert scales, ranging from 1 to 5. The overall score ranges from 0 (no regrets) to 100 (maximum regrets). Lower the score, lesser is the self-reported decisional regret.
  A Wilcoxon signed-rank test will be used. p-values < 0.05 will be considered statistically significant.
  The success of the study will be determined by a change in mean Decisional Regret Score in the intervention group by 11 points after 6-12 months of therapy initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Crowley, Principal Investigator — London Health Sciences Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Siyam T, Shahid A, Perram M, Zuna I, Haque F, Archundia-Herrera MC, Vohra S, Olson K. A scoping review of interventions to promote the adoption of shared decision-making (SDM) among health care professionals in clinical practice. Patient Educ Couns. 2019 Jun;102(6):1057-1066. doi: 10.1016/j.pec.2019.01.001. Epub 2019 Jan 3. PMID 30642716
- [Result] Briss P, Rimer B, Reilley B, Coates RC, Lee NC, Mullen P, Corso P, Hutchinson AB, Hiatt R, Kerner J, George P, White C, Gandhi N, Saraiya M, Breslow R, Isham G, Teutsch SM, Hinman AR, Lawrence R; Task Force on Community Preventive Services. Promoting informed decisions about cancer screening in communities and healthcare systems. Am J Prev Med. 2004 Jan;26(1):67-80. doi: 10.1016/j.amepre.2003.09.012. PMID 14700715
- [Result] Boland L, Graham ID, Legare F, Lewis K, Jull J, Shephard A, Lawson ML, Davis A, Yameogo A, Stacey D. Barriers and facilitators of pediatric shared decision-making: a systematic review. Implement Sci. 2019 Jan 18;14(1):7. doi: 10.1186/s13012-018-0851-5. PMID 30658670
- [Result] Lipstein EA, Lovell DJ, Denson LA, Kim SC, Spencer C, Ittenbach RF, Britto MT. High Levels of Decisional Conflict and Decision Regret When Making Decisions About Biologics. J Pediatr Gastroenterol Nutr. 2016 Dec;63(6):e176-e181. doi: 10.1097/MPG.0000000000001425. PMID 27749390
- [Result] O'Connor AM, Rostom A, Fiset V, Tetroe J, Entwistle V, Llewellyn-Thomas H, Holmes-Rovner M, Barry M, Jones J. Decision aids for patients facing health treatment or screening decisions: systematic review. BMJ. 1999 Sep 18;319(7212):731-4. doi: 10.1136/bmj.319.7212.731. PMID 10487995
- [Result] Shay LA, Lafata JE. Where is the evidence? A systematic review of shared decision making and patient outcomes. Med Decis Making. 2015 Jan;35(1):114-31. doi: 10.1177/0272989X14551638. Epub 2014 Oct 28. PMID 25351843
- [Result] Gravel K, Legare F, Graham ID. Barriers and facilitators to implementing shared decision-making in clinical practice: a systematic review of health professionals' perceptions. Implement Sci. 2006 Aug 9;1:16. doi: 10.1186/1748-5908-1-16. PMID 16899124
- [Result] Stacey D, Kryworuchko J, Bennett C, Murray MA, Mullan S, Legare F. Decision coaching to prepare patients for making health decisions: a systematic review of decision coaching in trials of patient decision AIDS. Med Decis Making. 2012 May-Jun;32(3):E22-33. doi: 10.1177/0272989X12443311. Epub 2012 Apr 13. PMID 22505617
- [Result] Lemberg DA, Day AS. Crohn disease and ulcerative colitis in children: an update for 2014. J Paediatr Child Health. 2015 Mar;51(3):266-70. doi: 10.1111/jpc.12685. Epub 2014 Jul 15. PMID 25039307
- [Result] Kappelman MD, Moore KR, Allen JK, Cook SF. Recent trends in the prevalence of Crohn's disease and ulcerative colitis in a commercially insured US population. Dig Dis Sci. 2013 Feb;58(2):519-25. doi: 10.1007/s10620-012-2371-5. Epub 2012 Aug 29. PMID 22926499
- [Result] Schildkraut V, Alex G, Cameron DJ, Hardikar W, Lipschitz B, Oliver MR, Simpson DM, Catto-Smith AG. Sixty-year study of incidence of childhood ulcerative colitis finds eleven-fold increase beginning in 1990s. Inflamm Bowel Dis. 2013 Jan;19(1):1-6. doi: 10.1002/ibd.22997. PMID 22532319
- [Result] Silva FA, Rodrigues BL, Ayrizono ML, Leal RF. The Immunological Basis of Inflammatory Bowel Disease. Gastroenterol Res Pract. 2016;2016:2097274. doi: 10.1155/2016/2097274. Epub 2016 Dec 14. PMID 28070181
- [Result] Walters TD, Kim MO, Denson LA, Griffiths AM, Dubinsky M, Markowitz J, Baldassano R, Crandall W, Rosh J, Pfefferkorn M, Otley A, Heyman MB, LeLeiko N, Baker S, Guthery SL, Evans J, Ziring D, Kellermayer R, Stephens M, Mack D, Oliva-Hemker M, Patel AS, Kirschner B, Moulton D, Cohen S, Kim S, Liu C, Essers J, Kugathasan S, Hyams JS; PRO-KIIDS Research Group. Increased effectiveness of early therapy with anti-tumor necrosis factor-alpha vs an immunomodulator in children with Crohn's disease. Gastroenterology. 2014 Feb;146(2):383-91. doi: 10.1053/j.gastro.2013.10.027. Epub 2013 Oct 23. PMID 24162032
- [Result] Forrest CB, Crandall WV, Bailey LC, Zhang P, Joffe MM, Colletti RB, Adler J, Baron HI, Berman J, del Rosario F, Grossman AB, Hoffenberg EJ, Israel EJ, Kim SC, Lightdale JR, Margolis PA, Marsolo K, Mehta DI, Milov DE, Patel AS, Tung J, Kappelman MD. Effectiveness of anti-TNFalpha for Crohn disease: research in a pediatric learning health system. Pediatrics. 2014 Jul;134(1):37-44. doi: 10.1542/peds.2013-4103. Epub 2014 Jun 16. PMID 24935993
- [Result] Hoentjen F, van Bodegraven AA. Safety of anti-tumor necrosis factor therapy in inflammatory bowel disease. World J Gastroenterol. 2009 May 7;15(17):2067-73. doi: 10.3748/wjg.15.2067. PMID 19418577
- [Result] Dulai PS, Thompson KD, Blunt HB, Dubinsky MC, Siegel CA. Risks of serious infection or lymphoma with anti-tumor necrosis factor therapy for pediatric inflammatory bowel disease: a systematic review. Clin Gastroenterol Hepatol. 2014 Sep;12(9):1443-51; quiz e88-9. doi: 10.1016/j.cgh.2014.01.021. Epub 2014 Jan 22. PMID 24462626
- [Result] Rosh JR, Turner D, Griffiths A, Cohen SA, Jacobstein D, Adedokun OJ, Padgett L, Terry NA, O'Brien C, Hyams JS. Ustekinumab in Paediatric Patients with Moderately to Severely Active Crohn's Disease: Pharmacokinetics, Safety, and Efficacy Results from UniStar, a Phase 1 Study. J Crohns Colitis. 2021 Nov 8;15(11):1931-1942. doi: 10.1093/ecco-jcc/jjab089. PMID 34037715
- [Result] Ledder O, Assa A, Levine A, Escher JC, de Ridder L, Ruemmele F, Shah N, Shaoul R, Wolters VM, Rodrigues A, Uhlig HH, Posovszky C, Kolho KL, Jakobsen C, Cohen S, Shouval DS, de Meij T, Martin-de-Carpi J, Richmond L, Bronsky J, Friedman M, Turner D. Vedolizumab in Paediatric Inflammatory Bowel Disease: A Retrospective Multi-Centre Experience From the Paediatric IBD Porto Group of ESPGHAN. J Crohns Colitis. 2017 Oct 1;11(10):1230-1237. doi: 10.1093/ecco-jcc/jjx082. PMID 28605483
- [Result] Grossi V, Lerer T, Griffiths A, LeLeiko N, Cabrera J, Otley A, Rick J, Mack D, Bousvaros A, Rosh J, Grossman A, Saeed S, Kay M, Boyle B, Oliva-Hemker M, Keljo D, Pfefferkorn M, Faubion W, Kappelman MD, Sudel B, Markowitz J, Hyams JS. Concomitant Use of Immunomodulators Affects the Durability of Infliximab Therapy in Children With Crohn's Disease. Clin Gastroenterol Hepatol. 2015 Oct;13(10):1748-56. doi: 10.1016/j.cgh.2015.04.010. Epub 2015 Apr 21. PMID 25911120
- [Result] De Bie CI, Hummel TZ, Kindermann A, Kokke FT, Damen GM, Kneepkens CM, Van Rheenen PF, Schweizer JJ, Hoekstra JH, Norbruis OF, Tjon A Ten WE, Vreugdenhil AC, Deckers-Kocken JM, Gijsbers CF, Escher JC, De Ridder L. The duration of effect of infliximab maintenance treatment in paediatric Crohn's disease is limited. Aliment Pharmacol Ther. 2011 Jan;33(2):243-50. doi: 10.1111/j.1365-2036.2010.04507.x. Epub 2010 Nov 14. PMID 21083595
- [Result] Schuler CL, Dodds C, Hommel KA, Ittenbach RF, Denson LA, Lipstein EA. Shared decision making in IBD: A novel approach to trial consent and timing. Contemp Clin Trials Commun. 2019 Sep 8;16:100447. doi: 10.1016/j.conctc.2019.100447. eCollection 2019 Dec. PMID 31538130
- [Result] Legare F, Kearing S, Clay K, Gagnon S, D'Amours D, Rousseau M, O'Connor A. Are you SURE?: Assessing patient decisional conflict with a 4-item screening test. Can Fam Physician. 2010 Aug;56(8):e308-14. PMID 20705870
- [Result] Bennett C, Graham ID, Kristjansson E, Kearing SA, Clay KF, O'Connor AM. Validation of a preparation for decision making scale. Patient Educ Couns. 2010 Jan;78(1):130-3. doi: 10.1016/j.pec.2009.05.012. Epub 2009 Jun 26. PMID 19560303
- [Result] Feenstra B, Lawson ML, Harrison D, Boland L, Stacey D. Decision coaching using the Ottawa family decision guide with parents and their children: a field testing study. BMC Med Inform Decis Mak. 2015 Feb 7;15:5. doi: 10.1186/s12911-014-0126-2. PMID 25889602
- See also: Ottawa Family Decision Guide © 2012 Lawson, Saarimaki, Kryworuchko, Boland, Feenstra, Stacey. Children's Hospital of Eastern Ontario Family Decision Services — https://decisionaid.ohri.ca/decguide.html
- See also: O'Connor AM. User Manual - Decisional Conflict Scale (16 item question format). Ottawa: Ottawa Hospital Research Institute; © 1993 [updated 2012]. 16 p. — http://decisionaid.ohri.ca/docs/develop/User_Manuals/UM_Decisional_Conflict.pdf
- See also: Graham ID, O'Connor AM. Preparation for Decision Making Scale; 2005 — http://decisionaid.ohri.ca/eval.html
- See also: O'Connor AM. User Manual - Decision Regret Scale. Ottawa: Ottawa Hospital Research Institute; © 1996 [modified 2003]. 3 p. — http://decisionaid.ohri.ca/docs/develop/User_Manuals/UM_Regret_Scale.pdf